CLINICAL TRIAL: NCT01355315
Title: Enhanced External Counterpulsation for Ischemic Cardiomyopathy
Brief Title: Enhanced External Counterpulsation
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shih-Hong Huang, Far Eastern Memorial Hospital
Other Study IDs: 95005; FEMH-95-C-039
Record Dates: First submitted 2008-06-18; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease; Congestive Heart Failure
Keywords: EECP; ischemic cardiomyopathy; endothelin-1; ischemia coronary artery diseases; congestive heart failure not amenable to standard procedures
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Enhanced external counterpulsation (EECP) is a noninvasive circulatory assist device that has been as a treatment option for refractory angina in left ventricular (LV) dysfunction. Recently, its potential role in heart failure management has been shown. However, although the concept of EECP was introduced almost four decades ago, and despite growing evidence supporting the clinical benefit and safety of this therapeutic modality, little is firmly established regarding the mechanisms responsible for the benefit of EECP include improvement in endothelial function, promotion of coronary collateralization, enhancement of ventricular function, and peripheral effects. Therefore, the major aim of this study is to provide an alternative treatment, EECP, for those unsuitable for standard procedures, especially for patients whose heart failure was caused by repeated myocardial infarction, called ischemic cardiomyopathy (ICMP), and to evaluate the clinical outcome and the endothelial function before and after 35 hours of EECP treatment.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria is left ventricular ejection fraction (LVEF) less than 40% by means of left ventricular angiography and symptomatic mild-to-moderate heart failure (New York Heart Association [NYHA] functional class II-III). The patient was included if there is no suitable target for either percutaneous coronary intervention or surgical bypass grafting.

Exclusion Criteria:

* IF he/she has moderate or severe aortic regurgitation (AR), history of deep vein thrombosis, or significant arrhythmia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ischemia coronary artery diseases and congestive heart failure not amenable to standard procedures
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual)